CLINICAL TRIAL: NCT01250379
Title: A Phase III Randomized Study Evaluating the Efficacy and Safety of Continued and Re-induced Bevacizumab in Combination With Chemotherapy for Patients With Locally Recurrent or Metastatic Breast Cancer After First-line Chemotherapy and Bevacizumab Treatment
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Chemotherapy in Patients With Breast Cancer Progressing After First-Line Therapy With Avastin and Chemotherapy (TANIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO22998; 2010-020998-16
Record Dates: First submitted 2010-11-25; First posted 2010-11-30 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Drug Therapy

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Chemotherapy
- 2 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Chemotherapy

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 10 mg/ kg iv every 2 weeks or 15 mg/kg iv every 3 weeks
  Arms: 2
Drug: Chemotherapy — Standard chemotherapy (doublets not allowed)

SUMMARY:
This randomized, open-label, parallel-group study will assess the efficacy and s afety of Avastin (bevacizumab) in combination with chemotherapy versus chemother apy alone as second- and third-line therapy in patients with locally recurrent o r metastatic breast cancer progressing after first-line therapy with Avastin and chemotherapy. Patients will be randomized to receive either Avastin (15 mg/kg e very 3 weeks or 10 mg/kg every 2 weeks intravenously) plus standard chemotherapy or chemotherapy alone. Anticipated time on study treatment is until third-line disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, >/= 18 years of age
* Histologically confirmed HER2-negative breast cancer
* Disease progression during or following first-line treatment with Avastin and chemotherapy for locally recurrent or metastatic breast cancer
* Avastin treatment in first-line setting must have been a minimum of 4 cycles (15 mg/kg) or 6 cycles (10 mg/kg) in combination with chemotherapy
* ECOG performance status 0-2
* At least 28 days since prior radiation therapy or surgery and recovery from treatment

Exclusion Criteria:

* Anti-angiogenic therapy or anti-vascular endothelial growth factors other than Avastin for first-line treatment
* Active malignancy other than superficial basal cell and superficial squamous cell carcinoma of the skin, or in situ carcinoma of the cervix or breast within the last 5 years
* Inadequate renal function
* Clinically relevant cardio-vascular disease
* Known CNS disease except for treated brain metastases
* Chronic daily treatment with high-dose aspirin (>325 mg/day) or clopidogrel (>75 mg/day)
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (117):
- Argentina (2):
  - Buenos Aires
  - San Miguel de Tucumán
- Austria (8):
  - Feldkirch
  - Graz
  - Innsbruck
  - Krems
  - Salzburg
  - Steyr
  - Vienna
  - Villach
- Brazil (3):
  - Goiânia, Goiás
  - Porto Alegre, Rio Grande do Sul
  - Itajaí, Santa Catarina
- Split, Croatia
- France (26):
  - Amiens
  - Angers
  - Besançon
  - Bordeaux
  - Boulogne-sur-Mer
  - Brest
  - Caen
  - Clermont-Ferrand
  - Dijon
  - Grenoble
  - Limoges
  - Marseille
  - Montpellier
  - Nancy
  - Nantes
  - Paris
  - Pierre-Bénite
  - Reims
  - Rouen
  - Saint-Cloud
  - Saint-Grégoire
  - Saint-Jean
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Strasbourg
  - Toulouse
- Germany (26):
  - Amberg
  - Aschaffenburg
  - Berlin
  - Bielefeld
  - Chemnitz
  - Cologne
  - Dresden
  - Düsseldorf
  - Essen
  - Freiburg im Breisgau
  - Göttingen
  - Hamburg
  - Hanover
  - Heidelberg
  - Karlsruhe
  - Mannheim
  - München
  - Münster
  - Naunhof
  - Neuss
  - Nordhausen
  - Osnabrück
  - Ravensburg
  - Stade
  - Stralsund
  - Wiesbaden
- Greece (4):
  - Athens
  - Ioannina
  - Pátrai
  - Thessaloniki
- Hungary (2):
  - Budapest
  - Szeged
- Israel (7):
  - Beersheba
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (15):
  - Cosenza, Calabria
  - Benevento, Campania
  - Napoli, Campania
  - Reggio Emilia, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Monza, Lombardy
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Macerata, The Marches
  - Florence, Tuscany
  - Pisa, Tuscany
  - Pontedera, Tuscany
  - Verona, Veneto
- Slovakia (5):
  - Bardejov
  - Bratislava
  - Košice
  - Nové Zámky
  - Prešov
- Spain (15):
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Santander, Cantabria
  - Castellon, Castellon
  - Córdoba, Cordoba
  - Donostia / San Sebastian, Guipuzcoa
  - León, Leon
  - Lleida, Lerida
  - Madrid, Madrid
  - Málaga, Malaga
  - Murcia, Murcia
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Switzerland (3):
  - Aarau
  - Chur
  - Zurich

REFERENCES:
- [Derived] Vrdoljak E, Marschner N, Zielinski C, Gligorov J, Cortes J, Puglisi F, Aapro M, Fallowfield L, Fontana A, Inbar M, Kahan Z, Welt A, Levy C, Brain E, Pivot X, Putzu C, Gonzalez Martin A, de Ducla S, Easton V, von Minckwitz G. Final results of the TANIA randomised phase III trial of bevacizumab after progression on first-line bevacizumab therapy for HER2-negative locally recurrent/metastatic breast cancer. Ann Oncol. 2016 Nov;27(11):2046-2052. doi: 10.1093/annonc/mdw316. Epub 2016 Aug 8. PMID 27502725
- [Derived] von Minckwitz G, Puglisi F, Cortes J, Vrdoljak E, Marschner N, Zielinski C, Villanueva C, Romieu G, Lang I, Ciruelos E, De Laurentiis M, Veyret C, de Ducla S, Freudensprung U, Srock S, Gligorov J. Bevacizumab plus chemotherapy versus chemotherapy alone as second-line treatment for patients with HER2-negative locally recurrent or metastatic breast cancer after first-line treatment with bevacizumab plus chemotherapy (TANIA): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1269-78. doi: 10.1016/S1470-2045(14)70439-5. Epub 2014 Sep 28. PMID 25273342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 556 participants were screened and of these, 494 were randomized.
Groups:
- Chemotherapy (CT) Arm: Participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site until disease progression, unacceptable toxicity, participant request for withdrawal, until the maximum cumulative dose of anthracycline was reached, or end of study (24 months after randomization of the last participant). Upon second-line disease progression participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site until disease progression, unacceptable toxicity, participant request for withdrawal, or end of study. Upon subsequent disease progression participants received treatment according the standard of care of the treatment site until end of study.
- Chemotherapy Plus Bevacizumab (CT+BV) Arm: Participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site plus bevacizumab, 15 milligrams per kilogram (mg/kg), intravenously (IV), every 3 weeks, or 10 mg/kg, IV, every 2 weeks until disease progression, unacceptable toxicity, participant request for withdrawal, until the maximum cumulative dose of anthracycline was reached, or end of study (24 months after randomization of the last participant). Upon second-line disease progression participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site plus bevacizumab, 15 mg/kg, IV, every 3 weeks, or 10 mg/kg, IV, every 2 weeks until disease progression, unacceptable toxicity, participant request for withdrawal, or end of study. Upon subsequent disease progression participants received treatment according the standard of care of the treatment site until end of study.
Period: Overall Study
Arm/Group | Chemotherapy (CT) Arm | Chemotherapy Plus Bevacizumab (CT+BV) Arm
Started | 247 | 247
Completed | 45 (Participants under study follow-up as of Data Cutoff 30 April 2015 were considered as completers.) | 54 (Participants under study follow-up as of Data Cutoff 30 April 2015 were considered as completers.)
Not Completed | 202 | 193
Not completed — Death | 141 | 148
Not completed — Withdrawal by Subject | 32 | 20
Not completed — Physician Decision | 11 | 3
Not completed — Protocol Violation | 2 | 8
Not completed — Lost to Follow-up | 9 | 6
Not completed — Adverse Event | 5 | 4
Not completed — Other | 0 | 4
Not completed — Participant noncompliance | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants.
Groups:
- CT Arm: Participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site until disease progression, unacceptable toxicity, participant request for withdrawal, until the maximum cumulative dose of anthracycline was reached, or end of study (24 months after randomization of the last participant). Upon second-line disease progression participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site until disease progression, unacceptable toxicity, participant request for withdrawal, or end of study. Upon subsequent disease progression participants received treatment according the standard of care of the treatment site until end of study.
- CT+BV Arm: Participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site plus bevacizumab, 15 mg/kg, IV, every 3 weeks, or 10 mg/kg, IV, every 2 weeks until disease progression, unacceptable toxicity, participant request for withdrawal, until the maximum cumulative dose of anthracycline was reached, or end of study (24 months after randomization of the last participant). Upon second-line disease progression participants received a single-agent chemotherapy at the discretion of the investigator according to the standard of care at the investigator's site plus bevacizumab, 15 mg/kg, IV, every 3 weeks, or 10 mg/kg, IV, every 2 weeks until disease progression, unacceptable toxicity, participant request for withdrawal, or end of study. Upon subsequent disease progression participants received treatment according the standard of care of the treatment site until end of study.
- Total: Total of all reporting groups
Arm/Group | CT Arm | CT+BV Arm | Total
Number analyzed (Participants) | 247 | 247 | 494
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.83) | 55.8 (11.17) | 55.2 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 247 | 494
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Second-Line Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1)
Description: Second-line PFS was defined as the time from randomization to progressive disease (PD) or death due to any cause during their second-line of treatment with bevacizumab and/or chemotherapy, whichever occurred first. For target lesions (TLs), PD was defined at least a 20 percent (%) increase in the sum of the largest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For non-target lesions (NTLs), PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without second-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: Baseline (less than or equal to [≤] 28 days after randomization), every 8-9 weeks thereafter according to the standard of care of the treatment site until approximately 3 years
Population: Intent-to-Treat (ITT) population - all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 88.7 | 93.9

2. Primary Outcome: Second-Line PFS
Description: The median time, in months, from randomization to second-line PFS event. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without second-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: Baseline (≤28 days after randomization), every 8-9 weeks thereafter according to the standard of care of the treatment site until approximately 3 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
months | 4.2 [3.9 to 5.3] | 6.3 [5.5 to 7.6]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.0204, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.97] — The 95% confidence interval (CI) was estimated using Cox proportional hazards methodology. The stratification factors used in the analysis were hormone receptor status, first-line PFS, choice of chemotherapy, and lactate dehydrogenase (LDH) level
Statistical Analysis 2: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.0245, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.67 to 0.97] — Unstratified analysis

3. Secondary Outcome: Second-Line PFS by Baseline Risk Factor (Data Cutoff 20 December 2013)
Description: The median time, in months, from randomization to second-line PFS event according to the following baseline risk factors: hormone receptor negative, HER2 negative (triple negative), hormone receptor positive/HER-2 negative (HR-pos/HER-neg), first-line PFS less than (<) 6 months, first-line PFS greater than or equal to (≥) 6 months, taxane chemotherapy (chemo), non-taxane chemo, vinorelbine chemo, LDH ≤ 1.5 upper limit of normal (ULN), LDH greater than (>) 1.5 ULN, < 65 years of age, ≥ 65 years of age, < 70 years of age, ≥ 70 years of age, < 3 metastatic organ sites, ≥ 3 metastatic organ sites, bevacizumab-free (B-free) interval ≤ 6 weeks, B-free > 6 weeks, disease-free (D-free) interval ≤ 24 months, D-free > 24 months, D-free ≤ 12 months, and D-free > 12 months. Participants without second-line PD or death were censored at the date of last tumor assessment where non-progression was documented. PD: defined in Outcome measure 1. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: ITT population. Here, Number of participants analyzed equals (=) participants evaluable for this outcome measure and number (n) = number of participants included in the analysis for the specified risk factor.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 226 | 219
months
  HR-neg (n=60,56) | 2.1 [2.0 to 3.9] | 4.9 [3.4 to 6.1]
  HR-pos/HER-neg (n=187,191) | 4.7 [4.2 to 6.2] | 6.7 [6.0 to 7.8]
  PFS <6 months (n=69,68) | 3.9 [2.3 to 4.3] | 5.1 [4.1 to 6.9]
  PFS ≥6 months (n=178,179) | 4.6 [3.9 to 6.1] | 6.4 [5.8 to 7.6]
  Taxane chemo (n=32,32) | 3.2 [1.7 to 5.3] | 6.9 [4.9 to 9.8]
  Non-taxane chemo (n=191,188) | 4.4 [3.9 to 5.8] | 6.0 [4.9 to 6.8]
  Vinorelbine chemo (n=24,27) | 2.4 [1.8 to 4.3] | 6.5 [4.2 to 11.1]
  LDH ≤ 1.5 ULN (n=207,210) | 4.4 [3.9 to 6.0] | 6.3 [5.5 to 7.6]
  LDH > 1.5 ULN (n=40,37) | 2.1 [1.7 to 3.9] | 5.8 [2.5 to 7.3]
  < 65 years of age (n=196,183) | 4.2 [3.9 to 4.7] | 6.1 [4.7 to 6.9]
  ≥ 65 years of age (n=51,64) | 4.2 [2.2 to 7.8] | 6.7 [5.5 to 8.0]
  < 70 years of age (n=226,219) | 4.2 [3.7 to 4.6] | 6.2 [5.3 to 7.3]
  ≥ 70 years of age (n=21,28) | 7.8 [2.2 to 11.9] | 6.7 [4.1 to 11.2]
  < 3 metastatic organ sites (n=158,167) | 4.2 [3.9 to 6.1] | 6.9 [6.0 to 8.2]
  ≥ 3 metastatic organ sites (n=88,80) | 4.0 [2.1 to 4.9] | 4.7 [4.1 to 6.2]
  B-free ≤ 6 weeks (n=165,149) | 4.2 [3.6 to 4.6] | 5.8 [4.4 to 6.6]
  B-free > 6 weeks (n=81,98) | 4.4 [3.3 to 6.3] | 7.6 [6.0 to 9.5]
  D-free ≤ 24 months (n=58,53) | 2.8 [2.0 to 3.9] | 5.8 [4.2 to 6.3]
  D-free > 24 months (n=138,156) | 4.9 [4.0 to 6.1] | 6.5 [5.5 to 8.1]
  D-free ≤ 12 months (n=24,18) | 2.1 [1.3 to 5.8] | 5.8 [3.9 to 9.7]
  D-free > 12 months (n=172,191) | 4.3 [3.9 to 5.7] | 6.3 [5.3 to 7.6]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: HR-neg; Test type: Superiority or Other; p = 0.0088, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.40 to 0.88]
Statistical Analysis 2: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: HR-pos/HER-neg; Test type: Superiority or Other; p = 0.1196, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.05]
Statistical Analysis 3: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: PFS <6 months; Test type: Superiority or Other; p = 0.0110, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.43 to 0.90]
Statistical Analysis 4: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: PFS ≥6 months; Test type: Superiority or Other; p = 0.0816, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.03]
Statistical Analysis 5: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: taxane chemo; Test type: Superiority or Other; p = 0.0395, Log Rank; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.31 to 0.98]
Statistical Analysis 6: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: non-taxane chemo; Test type: Superiority or Other; p = 0.1385, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.68 to 1.06]
Statistical Analysis 7: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: vinorelbine chemo; Test type: Superiority or Other; p = 0.0029, Log Rank; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.22 to 0.75]
Statistical Analysis 8: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: LDH ≤ 1.5 ULN; Test type: Superiority or Other; p = 0.0171, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.62 to 0.96]
Statistical Analysis 9: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: LDH > 1.5 ULN; Test type: Superiority or Other; p = 0.1797, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.46 to 1.16]
Statistical Analysis 10: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: < 65 years of age; Test type: Superiority or Other; p = 0.0229, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.62 to 0.97]
Statistical Analysis 11: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: ≥ 65 years of age; Test type: Superiority or Other; p = 0.2139, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.51 to 1.16]
Statistical Analysis 12: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: < 70 years of age; Test type: Superiority or Other; p = 0.0021, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.59 to 0.89]
Statistical Analysis 13: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: ≥ 70 years of age; Test type: Superiority or Other; p = 0.5216, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.64 to 2.39]
Statistical Analysis 14: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: < 3 metastatic organ sites; Test type: Superiority or Other; p = 0.0148, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.94]
Statistical Analysis 15: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: ≥ 3 metastatic organ sites; Test type: Superiority or Other; p = 0.3102, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.61 to 1.17]
Statistical Analysis 16: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: B-free ≤ 6 weeks; Test type: Superiority or Other; p = 0.0967, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.64 to 1.04]
Statistical Analysis 17: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: B-free > 6 weeks; Test type: Superiority or Other; p = 0.0489, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.51 to 1.00]
Statistical Analysis 18: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: D-free ≤ 24 months; Test type: Superiority or Other; p = 0.0176, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.41 to 0.92]
Statistical Analysis 19: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: D-free > 24 months; Test type: Superiority or Other; p = 0.2318, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.66 to 1.11]
Statistical Analysis 20: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: D-free ≤ 12 months; Test type: Superiority or Other; p = 0.0568, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.26 to 1.03]
Statistical Analysis 21: Comparison: CT Arm vs CT+BV Arm; Subgroup analysis: D-free > 12 months; Test type: Superiority or Other; p = 0.1143, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.66 to 1.05]

4. Secondary Outcome: Percentage of Participants With a Second-Line Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) According to RECIST v1.1 (Data Cutoff 20 December 2013)
Description: BOR was defined as a confirmed CR or PR during second-line treatment. For TLs, CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. The 95% Cl was determined using the Pearson-Clopper method.
Time Frame: as for outcome 2
Population: ITT population; only randomized participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 185 | 182
percentage of participants | 16.8 [11.7 to 22.9] | 20.9 [15.2 to 27.5]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.3457, Chi-squared; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-4.2 to 12.4] — The 95% CI was estimated using Hauck-Anderson methodology

5. Secondary Outcome: Percentage of Participants With a Second-Line CR, PR, Stable Disease, and PD According to RECIST v1.1 (Data Cutoff 20 December 2013)
Description: For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD; SD was defined as neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD; and PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels; stable disease was defined as the persistence of 1 or more NTLs and/or maintenance of tumor marker levels above normal limits; and PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. The 95% CI was determined using the Pearson-Clopper method.
Time Frame: as for outcome 2
Population: ITT population; only randomized participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 185 | 182
percentage of participants
  CR | 1.1 [0.1 to 3.9] | 0.5 [0.0 to 3.0]
  PR | 15.7 [10.8 to 21.7] | 20.3 [14.7 to 26.9]
  Stable disease | 33.5 [26.8 to 40.8] | 48.9 [41.4 to 56.4]
  PD | 41.1 [33.9 to 48.5] | 24.2 [18.1 to 31.1]
  Unable to assess | 8.6 [5.0 to 13.7] | 6.0 [3.1 to 10.6]

6. Secondary Outcome: Duration of Second-Line Objective Response (Data Cutoff 20 December 2013)
Description: The median time, in months, from the date of the first second-line documentation of CR or PR according to RECIST v1.1 to the date of the first second-line documentation of PD or death due to any cause. For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD; and PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels, and PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants with CR or PR who had experienced neither disease progression nor died were censored at the date of the last available tumor assessment when the participant was known to be progression free.
Time Frame: as for outcome 2
Population: ITT population; only randomized participants with a CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 31 | 38
months | 10.6 [4.4 to 16.7] | 8.3 [6.1 to 10.3]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.9825, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.51 to 1.99] — The 95% CI was estimated using Cox proportional hazards methodology. The stratification factors used in stratified analysis were hormone receptor status, first-line PFS, choice of chemotherapy, and LDH level
Statistical Analysis 2: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.3601, Log Rank; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.73 to 2.34] — Unstratified analysis

7. Secondary Outcome: Percentage of Participants With a Second-Line Documented CR or PR According to RECIST v1.1 Estimated to be Alive and Free of Disease Progression at Months 3, 6, and 9 (Data Cutoff 20 December 2013)
Description: Duration of objective response was defined as the median time, in months, from the date of the first second-line documentation of CR or PR to the date of the first second-line documentation of PD or death due to any cause. For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD; and PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels, and PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants with CR or PR who had experienced neither disease progression nor died were censored at the date of the last available tumor assessment when the participant was known to be progression free.
Time Frame: Months 3, 6, and 9
Population: ITT population; only randomized participants with a CR or PR were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 31 | 38
percentage of participants
  Month 3 | 96.7 [78.6 to 99.5] | 100.0 [NA to NA] — 95% CI data was not applicable (NA) because all participants were estimated to be alive and free of disease progression at this time point.
  Month 6 | 69.0 [48.9 to 82.5] | 72.8 [55.3 to 84.4]
  Month 9 | 60.9 [40.4 to 76.3] | 40.8 [24.6 to 56.3]

8. Secondary Outcome: Percentage of Participants With Third-Line PFS According to RECIST v1.1
Description: Third-line PFS was defined as the time from the date of first dose of third-line bevacizumab and/or chemotherapy to the date of third-line PD or death due to any cause. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without second-line PD or death were censored at the date of last tumor assessment where non-progression was documented. Participants without third-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: First dose of third-line treatment until PD or death due to any cause (assessed every 8-9 weeks, over a period of approximately 14 months)
Population: Third line ITT population: all randomized participants who received third-line treatment.
Measure: Number; unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 105 | 129
percentage of participants | 94.3 | 96.1

9. Secondary Outcome: Third-Line PFS
Description: The median time, in months, from the first dose of third-line bevacizumab and/or chemotherapy to third-line PD or death due to any cause. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without third-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: First dose of third-line treatment until PD or death due to any cause (over a period of approximately 14 months)
Population: Third line ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 105 | 129
months | 2.9 [2.2 to 3.9] | 3.8 [2.4 to 5.1]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.1080, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.59 to 1.06] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.0625, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.59 to 1.02] — Unstratified analysis

10. Secondary Outcome: Percentage of Participants With Second- and Third-Line PFS According to RECIST v1.1
Description: Second- and third-line PFS was defined as the time from the date randomization to the date of third-line PD or death due to any cause. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without third-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: Baseline (≤28 days after randomization), every 8-9 weeks thereafter according to the standard of care of the treatment site until approximately 4 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 71.7 | 83.4

11. Secondary Outcome: Second- and Third-Line PFS
Description: The median time, in months, from randomization to second-line and third-line PFS event. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without third-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: as for outcome 10
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
months | 10.7 [9.2 to 12.5] | 12.8 [10.7 to 14.5]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.1349, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.68 to 1.05] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.0863, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.68 to 1.03] — Unstratified analysis

12. Secondary Outcome: Percentage of Participants With Second- and Third-Line Tumor Progression
Description: Second- and third-line tumor progression was defined as occurrence of third-line PD according to RECIST v1.1 or death due to progression of disease. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without third-line PD or death due to progression of disease were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: as for outcome 10
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 67.2 | 75.3

13. Secondary Outcome: Time to Second- and Third-Line Tumor Progression
Description: The median time, in months, from randomization to second- and third-line tumor progression. Second- and third-line tumor progression was defined as third-line PD according to RECIST v1.1 or death due to progression of disease. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without third-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: as for outcome 10
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
months | 11.2 [9.4 to 12.7] | 13.3 [12.0 to 15.5]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.0744, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.65 to 1.02] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.0503, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 1.00] — Unstratified analysis

14. Primary Outcome: Percentage of Participants Estimated to be Alive and Free of Second-Line Disease Progression at Month 6
Description: Second-line PFS was defined as the time from randomization to PD or death due to any cause during their second-line of treatment with bevacizumab and/or chemotherapy, whichever occurred first. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without second-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: Month 6
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 40.7 [34.3 to 47.0] | 54.2 [47.7 to 60.3]

15. Secondary Outcome: Percentage of Participants Who Died
Description: Percentage of participants who died due to any reason were reported.
Time Frame: Baseline until death (up to approximately 4 years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 63.2 | 66.0

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the median time, in months, from the date of randomization to the date of death, due to any cause. Participants who had not died were censored at the date the patient was last known to be alive.
Time Frame: Baseline until death (up to approximately 4 years)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
months | 18.7 [15.4 to 21.2] | 19.7 [17.6 to 21.0]
Statistical Analysis 1: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.7253, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.76 to 1.21] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: CT Arm vs CT+BV Arm; Test type: Superiority or Other; p = 0.5332, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.75 to 1.16] — Unstratified analysis

17. Secondary Outcome: Percentage of Participants Estimated to be Surviving at Months 6, 12, 18, and 24
Description: OS was defined as the median time, in months, from the date of randomization to the date of death, due to any cause.
Time Frame: Months 6, 12, 18, and 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants
  Month 6 | 85.2 [79.9 to 89.2] | 90.4 [85.9 to 93.5]
  Month 12 | 68.6 [62.0 to 74.3] | 72.4 [66.2 to 77.7]
  Month 18 | 52.8 [46.0 to 59.3] | 54.9 [48.2 to 61.0]
  Month 24 | 38.4 [31.8 to 44.9] | 37.6 [31.3 to 43.9]

18. Secondary Outcome: Percentage of Participants Experiencing Problems by European Quality of Life Instrument (EQ-5D) Category (Data Cutoff 20 December 2013)
Description: The EQ-5D is composed of 5 single-item measures where participants responded to questions assessing health status by responding with either "no problems", "some problems", or "extreme problems" in the following categories: mobility (M) ("no problems"="I have no problems in walking about" to "extreme problems"="I am confined to bed"), self-care (SC) ("no problems"="I have no problems with self-care" to "extreme problems"="I am unable to wash or dress myself"), usual activities (UA) ("no problems"="I have no problems performing my usual activities" to "extreme problems"="I am unable to perform my usual activities"), pain/discomfort (P/D) ("no problems"="I have no pain or discomfort" to "extreme problems"="I have extreme pain or discomfort"), and anxiety/depression (A/D) ("no problems"="I am not anxious or depressed" to "extreme problems"='I am extremely anxious or depressed").
Time Frame: Baseline, during second-line treatment at Weeks 8 and 16 (4-week cycles) or Weeks 9 and 18 (3-week cycles) and at second-line PD (up to approximately 3 years)
Population: ITT population. Here, Number of participants analyzed = participants evaluable for this outcome measure and n=number of participants completing the questionnaires at the corresponding timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 214 | 224
percentage of participants
  BL: M, no problems (n=214,224) | 60.3 | 64.3
  BL: M, some problems (n=214,224) | 36.4 | 34.8
  BL: M, extreme problems (n=214,224) | 0.5 | 0.4
  BL: SC, no problems (n=214,224) | 82.7 | 85.7
  BL: SC, some problems (n=214,224) | 12.6 | 11.2
  BL: SC, extreme problems (n=214,224) | 0.5 | 1.8
  BL: UA, no problems (n=214,224) | 53.7 | 46.4
  BL: UA, some problems (n=214,224) | 40.2 | 48.7
  BL: UA, extreme problems (n=214,224) | 2.8 | 4.0
  BL: P/D, no problems (n=214,224) | 24.3 | 27.7
  BL: P/D, some problems (n=214,224) | 68.7 | 66.1
  BL: P/D, extreme problems (n=214,224) | 4.2 | 5.4
  BL: A/D, no problems (n=214,224) | 33.6 | 34.8
  BL: A/D, some problems (n=214,224) | 56.5 | 58.5
  BL: A/D, extreme problems (n=214,224) | 5.6 | 5.8
  Week 8/9: M, no problems (n=133,141) | 61.7 | 51.8
  Week 8/9: M, some problems (n=133,141) | 34.6 | 43.3
  Week 8/9: M, extreme problems (n=133,141) | 1.5 | 2.1
  Week 8/9: SC, no problems (n=133,141) | 82.0 | 75.9
  Week 8/9: SC, some problems (n=133,141) | 13.5 | 17.0
  Week 8/9: SC, extreme problems (n=133,141) | 1.5 | 3.5
  Week 8/9: UA, no problems (n=133,141) | 53.4 | 40.4
  Week 8/9: UA, some problems (n=133,141) | 40.6 | 51.8
  Week 8/9: UA, extreme problems (n=133,141) | 3.0 | 5.0
  Week 8/9: P/D, no problems (n=133,141) | 29.3 | 23.4
  Week 8/9: P/D, some problems (n=133,141) | 61.7 | 68.1
  Week 8/9: P/D, extreme problems (n=133,141) | 5.3 | 6.4
  Week 8/9: A/D, no problems (n=133,141) | 49.6 | 46.8
  Week 8/9: A/D, some problems (n=133,141) | 40.6 | 48.2
  Week 8/9: A/D, extreme problems (n=133,141) | 6.8 | 2.8
  Week 16/18: M, no problems (n=84,123) | 66.7 | 49.6
  Week 16/18: M, some problems (n=84,123) | 29.8 | 47.2
  Week 16/18: M, extreme problems (n=84,123) | 0.0 | 2.4
  Week 16/18: SC, no problems (n=84,123) | 81.0 | 78.9
  Week 16/18: SC, some problems (n=84,123) | 14.3 | 17.1
  Week 16/18: SC, extreme problems (n=84,123) | 0.0 | 3.3
  Week 16/18: UA, no problems (n=84,123) | 50.0 | 36.6
  Week 16/18: UA, some problems (n=84,123) | 42.9 | 56.1
  Week 16/18: UA, extreme problems (n=84,123) | 3.6 | 4.1
  Week 16/18: P/D, no problems (n=84,123) | 34.5 | 19.5
  Week 16/18: P/D, some problems (n=84,123) | 59.5 | 76.4
  Week 16/18: P/D, extreme problems (n=84,123) | 1.2 | 3.3
  Week 16/18: A/D, no problems (n=84,123) | 51.2 | 49.6
  Week 16/18: A/D, some problems (n=84,123) | 44.0 | 43.1
  Week 16/18: A/D, extreme problems (n=84,123) | 0.0 | 5.7
  Second-line PD: M, no problems (n=82,76) | 59.8 | 47.4
  Second-line PD: M, some problems (n=82,76) | 34.1 | 48.7
  Second-line PD: M, extreme problems (n=82,76) | 2.4 | 3.9
  Second-line PD: SC, no problems (n=82,76) | 76.8 | 75.0
  Second-line PD: SC, some problems (n=82,76) | 15.9 | 18.4
  Second-line PD: SC, extreme problems (n=82,76) | 1.2 | 6.6
  Second-line PD: UA, no problems (n=82,76) | 39.0 | 30.3
  Second-line PD: UA, some problems (n=82,76) | 50.0 | 59.2
  Second-line PD: UA, extreme problems (n=82,76) | 6.1 | 10.5
  Second-line PD: P/D, no problems (n=82,76) | 19.5 | 18.4
  Second-line PD: P/D, some problems (n=82,76) | 67.1 | 69.7
  Second-line PD: P/D, extreme problems (n=82,76) | 8.5 | 11.8
  Second-line PD: A/D, no problems (n=82,76) | 36.6 | 26.3
  Second-line PD: A/D, some problems (n=82,76) | 50.0 | 61.8
  Second-line PD: A/D, extreme problems (n=82,76) | 7.3 | 11.8

19. Secondary Outcome: Quality of Life Assessed As an Index Score Using the EQ-5D (Data Cutoff 20 December 2013)
Description: The EQ-5D is composed of 5 single-item measures where participants responded to questions assessing health status by responding with either "no problems", "some problems", or "extreme problems" in the following categories: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Based on large population surveys, an algorithm was used to combine the responses to each of these 5 measures into 1 single EQ-5D index score ranging from -0.59 (extreme problems) to +1 (no problems).
Time Frame: as for outcome 18
Population: ITT population. Here, Number of participants analyzed = participants evaluable for this outcome measure and n=number of participants who completed the assessment at the specified timepoint
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 202 | 219
score on a scale
  BL (n=202,219) | 0.6806 [0.6489 to 0.7122] | 0.6725 [0.6389 to 0.7061]
  Week 8/9 (n=127,135) | 0.6953 [0.6470 to 0.7437] | 0.6515 [0.6057 to 0.6973]
  Week 16/18 (n=80,118) | 0.7496 [0.7114 to 0.7879] | 0.6534 [0.6058 to 0.7010]
  Second-line PD (n=77,76) | 0.6290 [0.5642 to 0.6938] | 0.5553 [0.4736 to 0.6370]

20. Secondary Outcome: Change From Baseline in EQ-5D Index Scores (Data Cutoff 20 December 2013)
Description: The EQ-5D is composed of 5 single-item measures where participants responded to questions assessing health status by responding with either "no problems", "some problems", or "extreme problems" in the following categories: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Based on large population surveys, an algorithm was used to combine the responses to each of these 5 measures into 1 single EQ-5D index score ranging from -0.59 (extreme problems) to +1 (no problems) where a negative value indicated a worsening of perceived quality of life and a positive value indicated an improvement of perceived quality of life.
Time Frame: as for outcome 18
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 107 | 122
score on a scale
  Week 8/9 (n=107,122) | -0.0103 [-0.0482 to 0.0276] | -0.0370 [-0.0868 to 0.0127]
  Week 16/18 (n=68,110) | 0.0387 [-0.0025 to 0.0800] | -0.0508 [-0.1038 to 0.0021]
  Second-line PD (n=69,71) | -0.0884 [-0.1398 to -0.0371] | -0.0878 [-0.1649 to -0.0107]

21. Secondary Outcome: Quality of Life Assessed Using the EQ-5D Visual Analogue Scale (VAS) Scores (Data Cutoff 20 December 2013)
Description: The participant was asked to rate their overall health on a 0-100 millimeter (mm) vertical scale, where the lowest endpoint=0 (labeled as worst imaginable health state) and the highest endpoint =100 (labeled as the best imaginable health state). The participant marked the line corresponding to their assessment and the distance from the bottom was measured in millimeters. A higher value indicated a better health state.
Time Frame: as for outcome 18
Population: ITT population; n=number of participants who completed the assessment at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 200 | 212
mm
  BL (n=200,212) | 66.5 [64.1 to 69.0] | 63.4 [60.8 to 65.9]
  Week 8/9 (n=123,135) | 69.3 [66.4 to 72.1] | 66.5 [63.7 to 69.2]
  Week 16/18 (n=75,119) | 67.3 [63.3 to 71.3] | 66.4 [63.2 to 69.5]
  Second-line PD (n=78,75) | 63.7 [59.5 to 68.0] | 61.7 [57.0 to 66.5]

22. Secondary Outcome: Change From Baseline in VAS Scores (Data Cutoff 20 December 2013)
Description: The participant was asked to rate their overall health on a 0-100 mm vertical scale, where the lowest endpoint = 0 (labeled as worst imaginable health state) and the highest endpoint =100 (labeled as the best imaginable health state). The participant marked the line corresponding to their assessment and the distance from the bottom was measured in millimeters. A negative value indicated a worsening of perceived quality of life and a positive value indicated an improvement of perceived quality of life.
Time Frame: as for outcome 18
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 106 | 118
mm
  Week 8/9 (n=106,118) | -2.0 [-4.8 to 0.9] | 2.0 [-1.4 to 5.3]
  Week 16/18 (n=66,107) | -0.2 [-4.7 to 4.3] | 2.0 [-1.6 to 5.5]
  Second-line PD (n=70,69) | -5.1 [-9.1 to -1.0] | -1.3 [-5.5 to 3.0]

23. Secondary Outcome: Functional Assessment of Cancer Therapy-Breast (FACT-B) Scores (Data Cutoff 20 December 2013)
Description: The Functional Assessment of Cancer Therapy-Breast (FACT-B) is composed of 5 multi-item sections where participants responded to questions assessing symptoms (scale: 0-4; 0="not at all" and 4="very much"), as follows: physical well-being (PWB) (7 items, total score 0-28), social/family well-being (SWB) (7 items, total score 0-28), emotional well-being (EWB) (6 items, total score 0-24), functional well-being (FWB) (7 items, total score 0-28); and breast cancer score based on the additional concerns section of FACT-B (10 items, total score 0-40). The FACT-B Trial Outcomes Index (TOI) score=sum of PWB, FWB, and breast cancer score subscale scores (total score 0-96). The Functional Assessment of Cancer Therapy-General (FACT-G) total score=sum of PWB, SWB, EWB, and FWB subscales scores (total score 0-108). The FACT-B total score=sum of PWB, SWB, EWB, FWB, and breast cancer score subscales scores (total score 0-148). In all cases a higher value indicated a better perceived quality of life.
Time Frame: Baseline (≤28 days after randomization), every 8-9 weeks thereafter until second-line PD (up to approximately 3 years)
Population: ITT population. Here, Number of participants analyzed = participants evaluable for this outcome measure and n=number of participants who completed the questionnaire at the specified timepoints.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 215 | 224
score on a scale
  BL: PWB (n=215,222) | 20.621 [19.900 to 21.342] | 20.253 [19.500 to 21.006]
  BL: SWB (n=214,223) | 20.722 [20.028 to 21.416] | 20.674 [19.923 to 21.425]
  BL: EWB (n=215,224) | 14.847 [14.176 to 15.519] | 15.062 [14.419 to 15.704]
  BL: FWB (n=215,224) | 16.091 [15.289 to 16.894] | 15.726 [14.951 to 16.502]
  BL: Breast Cancer Score (n=210,224) | 24.986 [24.103 to 25.869] | 24.388 [23.578 to 25.198]
  BL: FACT-B TOI (n=204,219) | 61.677 [59.658 to 63.696] | 60.277 [58.365 to 62.189]
  BL: Total FACT-G Score (n=207,218) | 72.169 [69.919 to 74.419] | 71.864 [69.786 to 73.942]
  BL: Total FACT-B Score (n=201,218) | 96.908 [94.063 to 99.753] | 96.115 [93.485 to 98.746]
  Week 8/9: PWB (n=129,138) | 20.413 [19.413 to 21.413] | 19.156 [18.158 to 20.153]
  Week 8/9: SWB (n=127,135) | 20.833 [19.888 to 21.779] | 21.116 [20.245 to 21.987]
  Week 8/9: EWB (n=129,139) | 15.943 [15.070 to 16.815] | 16.671 [15.900 to 17.441]
  Week 8/9: FWB (n=129,139) | 16.662 [15.609 to 17.715] | 16.169 [15.180 to 17.158]
  Week 8/9: Breast Cancer Score (n=128,139) | 26.276 [25.188 to 27.364] | 25.884 [24.928 to 26.839]
  Week 8/9: FACT-B TOI (n=126,136) | 63.547 [60.975 to 66.118] | 61.279 [58.811 to 63.747]
  Week 8/9: Total FACT-G Score (n=122,134) | 74.255 [71.212 to 77.299] | 73.393 [70.603 to 76.184]
  Week 8/9: Total FACT-B Score (n=123,134) | 100.375 [96.582 to 104.169] | 99.213 [95.667 to 102.760]
  Week 16/18: PWB (n=83,107) | 21.733 [20.721 to 22.744] | 19.629 [18.571 to 20.688]
  Week 16/18: SWB (n=80,105) | 20.930 [19.855 to 22.006] | 20.843 [19.829 to 21.857]
  Week 16/18: EWB (n=80,107) | 17.330 [16.260 to 18.400] | 16.806 [15.961 to 17.650]
  Week 16/18: FWB (n=81,106) | 17.055 [15.818 to 18.291] | 15.920 [14.787 to 17.053]
  Week 16/18: Breast Cancer (n=81,106) | 26.923 [25.493 to 28.354] | 25.755 [24.630 to 26.880]
  Week 16/18: FACT-B TOI (n=78,105) | 65.628 [62.539 to 68.717] | 61.107 [58.309 to 63.905]
  Week 16/18: Total FACT-G (n=78,102) | 76.794 [73.269 to 80.318] | 73.269 [70.116 to 76.421]
  Week 16/18: Total FACT-B (n=76,103) | 103.503 [98.819 to 108.187] | 98.906 [94.865 to 102.948]
  Week 24/27: PWB (n=48,80) | 21.940 [20.599 to 23.282] | 18.965 [17.515 to 20.416]
  Week 24/27: SWB (n=47,78) | 20.840 [19.468 to 22.211] | 21.399 [20.192 to 22.606]
  Week 24/27: EWB (n=45,78) | 17.098 [15.719 to 18.477] | 16.438 [15.411 to 17.436]
  Week 24/27: FWB (n=45,79) | 18.244 [16.754 to 19.734] | 16.051 [14.861 to 17.241]
  Week 24/27: Breast Cancer (n=46,79) | 26.067 [24.146 to 27.988] | 24.632 [23.231 to 26.033]
  Week 24/27: FACT-B TOI (n=44,77) | 65.882 [61.991 to 69.653] | 60.014 [56.548 to 63.480]
  Week 24/27: Total FACT-G (n=44,77) | 78.305 [74.166 to 82.443] | 73.083 [69.365 to 76.801]
  Week 24/27: Total FACT-B (n=43,77) | 104.011 [98.433 to 109.588] | 97.795 [92.995 to 102.595]
  Week 32/36: PWB (n=26,44) | 22.949 [21.427 to 24.471] | 19.686 [18.121 to 21.250]
  Week 32/36: SWB (n=25,43) | 22.140 [20.433 to 23.847] | 21.222 [19.645 to 22.798]
  Week 32/36: EWB (n=26,44) | 18.385 [16.690 to 20.079] | 16.755 [15.481 to 18.028]
  Week 32/36: FWB (n=26,44) | 19.615 [17.875 to 21.356] | 17.195 [15.585 to 18.805]
  Week 32/36: Breast Cancer (n=26,43) | 29.568 [27.722 to 31.415] | 26.163 [24.457 to 27.869]
  Week 32/36: FACT-B TOI (n=26,42) | 72.132 [68.549 to 75.716] | 63.017 [59.199 to 66.836]
  Week 32/36: Total FACT-G (n=25,42) | 83.087 [78.178 to 87.995] | 74.879 [70.566 to 79.191]
  Week 32/36: Total FACT-B (n=25,42) | 112.904 [107.315 to 118.494] | 100.904 [95.302 to 106.506]
  Week 40/45: PWB (n=20,27) | 22.215 [20.583 to 23.847] | 20.630 [18.820 to 22.440]
  Week 40/45: SWB (n=21,26) | 19.658 [17.955 to 21.361] | 20.915 [19.146 to 22.685]
  Week 40/45: EWB (n=20,27) | 17.560 [15.708 to 19.412] | 16.067 [13.875 to 18.259]
  Week 40/45: FWB (n=20,27) | 18.450 [16.120 to 20.780] | 16.519 [13.901 to 19.136]
  Week 40/45: Breast Cancer (n=21,27) | 29.386 [27.156 to 31.616] | 23.819 [21.013 to 26.625]
  Week 40/45: FACT-B TOI (n=19,27) | 68.750 [63.981 to 73.518] | 60.967 [55.065 to 66.870]
  Week 40/45: Total FACT-G (n=19,26) | 76.955 [71.480 to 82.430] | 75.235 [68.901 to 81.568]
  Week 40/45: Total FACT-B (n=19,26) | 105.540 [98.512 to 112.568] | 99.072 [90.613 to 107.531]
  Week 48/54: PWB (n=13,24) | 23.308 [21.283 to 25.333] | 20.033 [18.124 to 21.943]
  Week 48/54: SWB (n=13,23) | 20.740 [18.953 to 22.527] | 20.450 [18.310 to 22.590]
  Week 48/54: EWB (n=13,23) | 19.308 [17.522 to 21.093] | 17.270 [15.494 to 19.045]
  Week 48/54: FWB (n=13,23) | 18.538 [16.586 to 20.491] | 16.268 [13.949 to 18.587]
  Week 48/54: Breast Cancer (n=13,23) | 28.912 [26.879 to 30.945] | 26.237 [22.842 to 29.632]
  Week 48/54: Fact-B TOI (n=13,23) | 70.758 [66.403 to 75.114] | 62.679 [55.941 to 69.418]
  Week 48/54: Total FACT-G (n=13,23) | 81.894 [76.424 to 87.363] | 74.162 [67.865 to 80.458]
  Week 48/54: Total FACT-B (n=13,23) | 110.806 [104.704 to 116.908] | 100.399 [91.294 to 109.503]
  Week 56/63: PWB (n=8,14) | 21.792 [18.958 to 24.626] | 20.298 [17.412 to 23.184]
  Week 56/63: SWB (n=8,14) | 19.583 [15.598 to 23.569] | 20.817 [17.629 to 24.004]
  Week 56/63: EWB (n=7,14) | 17.143 [13.389 to 20.897] | 15.714 [12.606 to 18.823]
  Week 56/63: FWB (n=7,14) | 17.143 [13.876 to 20.410] | 16.476 [12.633 to 20.319]
  Week 56/63: Breast Cancer (n=8,14) | 28.240 [23.931 to 32.548] | 25.459 [21.407 to 29.512]
  Week 56/63: FACT-B TOI (n=7,14) | 66.179 [55.888 to 76.469] | 62.233 [53.524 to 70.942]
  Week 56/63: Total FACT-G (n=6,14) | 73.667 [58.381 to 88.952] | 73.305 [62.863 to 83.746]
  Week 56/63: Total FACT-B (n=6,14) | 101.042 [81.841 to 120.242] | 98.764 [85.368 to 112.160]
  Week 64/72: PWB (n=7,9) | 21.857 [17.376 to 26.338] | 21.889 [19.569 to 24.209]
  Week 64/72: SWB (n=7,9) | 18.976 [16.352 to 21.600] | 22.685 [19.417 to 25.953]
  Week 64/72: EWB (n=7,9) | 18.143 [13.758 to 22.527] | 17.889 [14.274 to 21.503]
  Week 64/72: FWB (n=7,9) | 18.429 [14.658 to 22.199] | 16.037 [12.890 to 19.184]
  Week 64/72: Breast Cancer (n=7,9) | 27.464 [22.941 to 31.988] | 26.889 [22.584 to 31.194]
  Week 64/72: FACT-B TOI (n=7,9) | 67.750 [56.306 to 79.194] | 64.815 [56.516 to 73.114]
  Week 64/72: Total FACT-G (n=7,9) | 77.405 [63.847 to 90.963] | 78.500 [68.852 to 88.148]
  Week 64/72: Total FACT-B (n=7,9) | 104.869 [87.586 to 122.152] | 105.389 [92.415 to 118.363]
  Week 72/81: PWB (n=6,7) | 23.083 [18.906 to 27.260] | 21.000 [16.407 to 25.593]
  Week 72/81: SWB (n=5,7) | 19.667 [16.238 to 23.095] | 20.043 [14.019 to 26.067]
  Week 72/81: EWB (n=6,7) | 17.500 [13.476 to 21.524] | 18.114 [14.130 to 22.098]
  Week 72/81: FWB (n=6,7) | 17.333 [14.316 to 20.351] | 16.429 [11.339 to 21.518]
  Week 72/81: Breast Cancer (n=6,6) | 28.597 [24.421 to 32.774] | 25.333 [20.250 to 30.417]
  Week 72/81: FACT-B TOI (n=6,6) | 69.014 [59.566 to 78.462] | 60.833 [47.031 to 74.635]
  Week 72/81: Total FACT-G (n=5,7) | 76.467 [62.045 to 90.889] | 75.586 [57.141 to 94.030]
  Week 72/81: Total FACT-B (n=5,6) | 106.117 [88.146 to 124.087] | 97.211 [73.196 to 121.226]
  Week 80/90: PWB (n=2,3) | 19.250 [-32.634 to 71.134] | 18.000 [2.487 to 33.513]
  Week 80/90: SWB (n=2,3) | 18.375 [7.257 to 29.493] | 19.944 [3.434 to 36.455]
  Week 80/90: EWB (n=2,3) | 14.000 [-49.531 to 77.531] | 15.733 [-3.285 to 34.752]
  Week 80/90: FWB (n=2,3) | 15.000 [-35.825 to 65.825] | 12.333 [-1.348 to 26.015]
  Week 80/90: Breast Cancer (n=2,3) | 21.667 [0.490 to 42.844] | 25.000 [14.172 to 35.828]
  Week 80/90: FACT-B TOI (n=2,3) | 55.917 [-67.969 to 179.802] | 55.333 [20.085 to 90.581]
  Week 80/90: Total FACT-G (n=2,3) | 66.625 [-110.732 to 243.982] | 66.011 [2.191 to 129.831]
  Week 80/90: Total FACT-B (n=2,3) | 88.292 [-110.243 to 286.826] | 91.011 [20.313 to 161.709]
  Week 88/99: PWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 22.000 [NA to NA] — Standard deviation (SD) not calculated as only 1 participant was analyzed.
  Week 88/99: SWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 23.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: EWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 20.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: FWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 21.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: Breast Cancer (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 35.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: FACT-B TOI (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 78.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: Total FACT-G (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 86.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: Total FACT-B (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 121.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: PWB (n=2,1) | 26.000 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 22.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: SWB (n=2,1) | 24.383 [-3.782 to 52.549] | 21.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: EWB (n=2,2) | 22.000 [9.294 to 34.706] | 18.000 [-7.412 to 43.412]
  Week 96/108: FWB (n=2,2) | 21.083 [7.318 to 34.848] | 10.500 [-46.678 to 67.678]
  Week 96/108: Breast Cancer (n=2,2) | 30.389 [-2.788 to 63.566] | 24.500 [-7.266 to 56.266]
  Week 96/108: FACT-B TOI (n=2,1) | 77.472 [58.060 to 96.884] | 59.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: Total FACT-G (n=2,1) | 93.467 [38.830 to 148.103] | 74.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: Total FACT-B (n=2,1) | 123.856 [102.396 to 145.315] | 96.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 104/117: PWB (n=1,3) | 27.000 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 21.333 [17.539 to 25.128]
  Week 104/117: SWB (n=1,2) | 26.600 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 20.5000 [14.147 to 26.853]
  Week 104/117: EWB (n=1,3) | 22.000 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 18.000 [6.616 to 29.384]
  Week 104/117: FWB (n=1,3) | 22.000 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 11.000 [-1.908 to 23.908]
  Week 104/117: Breast Cancer (n=1,3) | 27.143 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 28.000 [19.395 to 36.605]
  Week 104/117: FACT-B TOI (n=1,3) | 76.143 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 60.333 [45.778 to 74.889]
  Week 104/117: Total FACT-G (n=1,2) | 97.600 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 70.500 [-50.209 to 191.209]
  Week 104/117: Total FACT-B (n=1,2) | 124.743 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 100.500 [-20.209 to 221.209]
  Week 112/126: PWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 14.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: SWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 15.400 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: EWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 15.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: FWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 11.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: Breast Cancer (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 20.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: FACT-B TOI (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 45.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: Total FACT-G (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 55.400 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: Total FACT-B (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 75.400 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Second-Line PD: PWB (n=89,81) | 19.086 [17.873 to 20.299] | 17.412 [15.977 to 18.846]
  Second-Line PD: SWB (n=88,79) | 20.623 [19.456 to 21.790] | 21.487 [20.335 to 22.639]
  Second-Line PD: EWB (n=88,80) | 15.111 [14.102 to 16.121] | 14.175 [12.872 to 15.478]
  Second-Line PD: FWB (n=88,80) | 15.447 [14.122 to 16.772] | 15.235 [13.877 to 16.593]
  Second-Line PD: Breast Cancer (n=85,81) | 24.978 [23.602 to 26.354] | 24.445 [22.989 to 25.901]
  Second-Line PD: FACT-B TOI (n=84,80) | 59.230 [56.033 to 62.428] | 57.002 [53.234 to 60.770]
  Second-Line PD: Total FACT-G (n=86,78) | 69.829 [66.264 to 73.393] | 68.485 [64.384 to 72.586]
  Second-Line PD: Total FACT-B (n=82,78) | 94.930 [90.240 to 99.619] | 92.983 [87.645 to 98.320]

24. Secondary Outcome: Change From Baseline in FACT-B Scores (Data Cutoff 20 December 2013)
Description: The FACT-B is composed of 5 multi-item sections where participants responded to questions assessing symptoms (scale: 0-4; 0="not at all" and 4="very much"), as follows: PWB (7 items, total score 0-28), SWB (7 items, total score 0-28), EWB (6 items, total score 0-24), FWB (7 items, total score 0-28); and breast cancer score based on the additional concerns section of FACT-B (10 items, total score 0-40). The FACT-B TOI score=sum of PWB, FWB, and breast cancer score subscale scores (total score 0-96). The FACT-G total score=sum of PWB, SWB, EWB, and FWB subscales scores (total score 0-108). The FACT-B total score=sum of PWB, SWB, EWB, FWB, and breast cancer score subscale scores (total score 0-148). In all cases a higher value indicated a better perceived quality of life.
Time Frame: Baseline (≤28 days after randomization), every 8-9 weeks thereafter until second-line PD (up to approximately 3 years)
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 118 | 128
score on a scale
  Week 8/9: PWB (n=118,125) | -1.281 [-2.219 to -0.344] | -1.289 [-2.239 to -0.338]
  Week 8/9: SWB (n=116,125) | 0.356 [-0.283 to 0.994] | 0.707 [-0.226 to 1.640]
  Week 8/9: EWB (n=116,128) | 0.408 [-0.274 to 1.089] | 1.024 [0.314 to 1.734]
  Week 8/9: FWB (n=117,128) | -0.226 [-1.043 to 0.591] | -0.240 [-1.027 to 0.548]
  Week 8/9: Breast Cancer Score (n=113,128) | 0.228 [-0.659 to 1.116] | 0.950 [0.121 to 1.780]
  Week 8/9: FACT-B TOI (n=110,122) | -1.361 [-3.295 to 0.573] | -0.357 [-2.407 to 1.693]
  Week 8/9: Total FACT-G Score (n=110,122) | -0.760 [-2.920 to 1.399] | 0.369 [-1.945 to 2.684]
  Week 8/9: Total FACT-B Score (n=108,120) | -0.728 [-3.332 to 1.876] | 1.342 [-1.544 to 4.229]
  Week 16/18: PWB (n=77,97) | 0.294 [-0,733 to 1.322] | -1.823 [-2.871 to -0.775]
  Week 16/18: SWB (n=74,97) | -0.443 [-1.411 to 0.525] | 0.359 [-0.678 to 1.397]
  Week 16/18: EWB (n=73,98) | 1.197 [0.415 to 1.979] | 0.921 [0.186 to 1.657]
  Week 16/18: FWB (n=75,98) | -0.548 [-1.666 to 0.570] | -0.517 [-1.422 to 0.389]
  Week 16/18: Breast Cancer (n=72,97) | 0.578 [-0.658 to 1.815] | 0.546 [-0.423 to 1.514]
  Week 16/18: FACT-TOI (n=68,95) | -0.483 [-3.149 to 2.183] | -1.732 [-4.049 to 0.586]
  Week 16/18: Total FACT-G (n=71,93) | -0.019 [-2.970 to 2.931] | -0.836 [-3.494 to 1.821]
  Week 16/18: Total Fact-B (n=66,93) | -0.007 [-3.744 to 3.730] | -0.127 [-3.421 to 3.167]
  Week 24/27: PWB (n=44,73) | 0.181 [-1.236 to 1.598] | -1.996 [-3.306 to -0.685]
  Week 24/27: SWB (n=44,72) | -0.193 [-1.490 to 1.104] | 1.375 [-0.001 to 2.750]
  Week 24/27: EWB (n=42,72) | 0.867 [-0.101 to 1.834] | 1.217 [0.366 to 2.067]
  Week 24/27: FWB (n=42,72) | 0.119 [-1.405 to 1.643] | 0.056 [-1.053 to 1.166]
  Week 24/27: Breast Cancer (n=40,72) | -0.038 [-1.723 to 1.647] | 0.078 [-1.106 to 1.262]
  Week 24/27: FACT-B TOI (n=38,70) | 0.221 [-3.411 to 3.853] | -1.573 [-4.383 to 1.238]
  Week 24/27: Total FACT-G (n=40,70) | 0.764 [-3.066 to 4.595] | 0.817 [-2.497 to 4.131]
  Week 24/27: Total FACT-B (n=37,70) | 0.793 [-4.106 to 5.693] | 1.157 [-2.828 to 5.142]
  Week 32/36: PWB (n=25,39) | 0.880 [-0.913 to 2.673] | -1.235 [-2.799 to 0.329]
  Week 32/36: SWB (n=24,40) | -0.388 [-1.754 to 0.979] | 1.036 [-1.209 to 3.281]
  Week 32/36: EWB (n=25,40) | 1.064 [-0.298 to 2.426] | 1.555 [0.204 to 2.906]
  Week 32/36: FWB (n=25,40) | 1.380 [-0.103 to 2.863] | 1.635 [-0.201 to 3.471]
  Week 32/36: Breast Cancer (n=23,40) | 0.928 [-1.916 to 3.771] | 1.278 [-0.435 to 2.990]
  Week 32/36: FACT-B TOI (n=23,38) | 3.123 [-1.390 to 7.637] | 1.471 [-2.522 to 5.464]
  Week 32/36: Total FACT-G (n=24,39) | 2.617 [-1.313 to 6.547] | 3.197 [-1.346 to 7.740]
  Week 32/36: Total FACT-B (n=22,38) | 3.529 [-2.074 to 9.132] | 3.896 [-1.579 to 9.370]
  Week 40/45: PWB (n=18,25) | 0.137 [-2.051 to 2.325] | -0.680 [-2.930 to 1.570]
  Week 40/45: SWB (n=19,24) | -0.589 [-2.436 to 1.259] | 0.951 [-1.590 to 3.492]
  Week 40/45: EWB (n=18,25) | 0.200 [-1.598 to 1.998] | 1.048 [-0.658 to 2.754]
  Week 40/45: FWB (n=18,25) | 1.417 [-0.562 to 3.395] | 0.857 [-0.893 to 2.608]
  Week 40/45: Breast Cancer (n=18,25) | 1.395 [-1.268 to 4.058] | 0.444 [-2.358 to 3.247]
  Week 40/45: FACT-B TOI (n=16,25) | 2.432 [-2.496 to 7.360] | 0.622 [-4.688 to 5.932]
  Week 40/45: Total FACT-G (n=17,24) | 1.444 [-3.342 to 6.231] | 2.432 [-3.035 to 7.899]
  Week 40/45: Total FACT-B (n=16,24) | 1.916 [-3.950 to 7.782] | 2.673 [-4.258 to 9.603]
  Week 48/54: PWB (n=13,20) | 1.295 [-2.037 to 4.627] | -1.833 [-3.721 to 0.055]
  Week 48/54: SWB (n=13,20) | 1.529 [-0.316 to 3.375] | 2.008 [-1.083 to 5.099]
  Week 48/54: EWB (n=13,20) | 1.492 [0.492 to 2.492] | 1.710 [-0.183 to 3.603]
  Week 48/54: FWB (n=13,20) | 2.269 [0.174 to 4.365] | 1.592 [-0.872 to 4.055]
  Week 48/54: Breast Cancer (n=12,20) | 0.599 [-1.714 to 2.912] | 1.897 [-0.463 to 4.258]
  Week 48/54: FACT-B TOI (n=12,20) | 4.044 [-2.832 to 10.919] | 1.656 [-3.691 to 7.002]
  Week 48/54: Total FACT-G (n=13,20) | 6.586 [1.392 to 11.780] | 3.477 [-2.596 to 9.550]
  Week 48/54: Total FACT-B (n=12,20) | 7.067 [0.241 to 13.894] | 5.374 [-2.391 to 13.139]
  Week 56/63: PWB (n=8,13) | -2.063 [-6.094 to 1.969] | -0.526 [-3.996 to 2.944]
  Week 56/63: SWB (n=8,13) | -1.500 [-5.699 to 2.699] | 3.033 [-1.729 to 7.796]
  Week 56/63: EWB (n=7,13) | 0.857 [-2.781 to 4.495] | 0.954 [-2.190 to 4.097]
  Week 56/63: FWB (n=7,13) | 0.000 [-4.835 to 4.835] | 5.654 [0.511 to 10.797]
  Week 56/63: Breast Cancer (n=8,13) | -0.830 [-6.133 to 4.474] | 1.675 [-1.291 to 4.641]
  Week 56/63: FACT-B TOI (n=7,13) | -3.591 [-17.803 to 10.621] | 6.803 [1.093 to 14.699]
  Week 56/63: Total FACT-G (n=6,13) | -4.083 [-22.930 to 14.764] | 9.115 [-3.820 to 22.050]
  Week 56/63: Total FACT-B (n=6,13) | -5.301 [-29.740 to 19.138] | 10.791 [-3.114 to 24.695]
  Week 64/72: PWB (n=7,9) | 0.000 [-6.733 to 6.733] | 0.926 [-1.491 to 3.342]
  Week 64/72: SWB (n=7,9) | -2.014 [-5.182 to 1.154] | 3.570 [-1.034 to 8.174]
  Week 64/72: EWB (n=7,9) | -0.057 [-3.537 to 3.423] | 3.667 [-0.630 to 7.964]
  Week 64/72: FWB (n=7,9) | 0.214 [-4.531 to 4.959] | 3.222 [-2.143 to 8.588]
  Week 64/72: Breast Cancer (n=7,9) | -2.298 [-7.507 to 2.912] | 3.086 [-1.361 to 7.534]
  Week 64/72: FACT-B TOI (n=7,9) | -2.083 [-17.130 to 12.963] | 7.235 [-3.624 to 18.093]
  Week 64/72: Total FACT-G (n=7,9) | -1.857 [-17.855 to 14.140] | 11.385 [-3.116 to 25.886]
  Week 64/72: Total FACT-B (n=7,9) | -4.155 [-24.302 to 15.993] | 14.472 [-4.192 to 33.135]
  Week 72/81: PWB (n=5,7) | 2.133 [-6.045 to 10.311] | -0.429 [-3.965 to 3.108]
  Week 72/81: SWB (n=4,7) | -1.208 [-5.126 to 2.710] | 6.829 [-3.189 to 16.846]
  Week 72/81: EWB (n=5,7) | -0.600 [-5.042 to 3.842] | 4.686 [-0.608 to 9.979]
  Week 72/81: FWB (n=5,7) | 0.000 [-5.341 to 5.341] | 7.381 [-1.169 to 15.931]
  Week 72/81: Breast Cancer (n=5,6) | -0.461 [-6.531 to 5.609] | 3.667 [-3.410 to 10.743]
  Week 72/81: FACT-B TOI (n=5,6) | 1.672 [-12.563 to 15.907] | 8.278 [-7.450 to 24.005]
  Week 72/81: Total FACT-G (n=4,7) | -0.167 [-22.161 to 21.828] | 18.467 [-1.867 to 38.801]
  Week 72/81: Total FACT-B (n=4,6) | 1.174 [-23.085 to 25.432] | 16.906 [-9.207 to 43.018]
  Week 80/90: PWB (n=2,3) | -3.750 [-30.221 to 22.721] | -3.000 [-11.605 to 5.605]
  Week 80/90: SWB (n=2,3) | -0.875 [-34.229 to 32.479] | 7.344 [-9.614 to 24.303]
  Week 80/90: EWB (n=2,3) | -4.000 [-42.119 to 34.119] | 4.733 [-18.466 to 27.932]
  Week 80/90: FWB (n=2,3) | -1.000 [-64.531 to 62.531] | 2.556 [-9.165 to 14.276]
  Week 80/90: Breast Cancer (n=2,3) | -5.833 [-29.128 to 17.461] | 3.667 [-11.512 to 18.845]
  Week 80/90: FACT-B TOI (n=2,3) | -10.583 [-77.291 to 56.124] | 3.222 [-30.212 to 36.657]
  Week 80/90: Total FACT-G (n=2,3) | -9.625 [-171.100 to 151.850] | 11.633 [-41.554 to 64.821]
  Week 80/90: Total FACT-B (n=2,3) | -15.458 [-153.638 to 122.722] | 15.300 [-48.177 to 78.777]
  Week 88/99: PWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -6.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: SWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 23.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: EWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 0.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: FWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 21.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: Breast Cancer (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 3.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: FACT TOI (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 18.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: Total FACT-G (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 38.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 88/99: Total FACT-B (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 41.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: PWB (n=2,1) | 7.333 [-51.962 to 66.629] | -3.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: SWB (n=2,1) | 2.183 [-23.441 to 27.808] | 1.400 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: EWB (n=2,1) | 0.000 [-12.706 to 12.706] | 6.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: FWB (n=2,1) | 6.583 [-13.535 to 26.701] | -1.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: Breast Cancer (n=2,1) | 3.167 [-41.305 to 47.638] | -3.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: FACT-B TOI (n=2,1) | 17.083 [11.789 to 22.378] | -7.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: Total FACT-G (n=2,1) | 16.100 [15.253 to 16.947] | 3.067 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 96/108: Total FACT-B (n=2,1) | 19.267 [-24.358 to 62.891] | 0.067 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 104/117: PWB (n=1,2) | 3.667 [NA to NA] — SD not calculated as only 1 participant was analyzed. | -2.000 [-40.119 to 36.119]
  Week 104/117: SWB (n=1,1) | 4.200 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 8.800 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 104/117: EWB (n=1,2) | 0.000 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 10.000 [-28.119 to 48.119]
  Week 104/117: FWB (n=1,2) | 8.000 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 2.333 [-56.962 to 61.629]
  Week 104/117: Breast Cancer (n=1,2) | 6.032 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 4.000 [-59.531 to 67.531]
  Week 104/117: FACT-B TOI (n=1,2) | 17.698 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 4.333 [-156.612 to 165.279]
  Week 104/117: Total FACT-G (n=1,1) | 15.867 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 29.800 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 104/117: Total GACT-B (n=1,1) | 21.898 [NA to NA] — SD not calculated as only 1 participant was analyzed. | 38.800 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: PWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -11.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: SWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -4.200 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: EWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | 5.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: FWB (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -5.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: Breast Cancer (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -5.000 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: FACT-B TOI (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -21.333 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: Total FACT-G (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -15.533 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Week 112/126: Total FACT-B (n=0,1) | NA [NA to NA] — Zero participants analyzed. | -20.533 [NA to NA] — SD not calculated as only 1 participant was analyzed.
  Second-Line PD: PWB (n=81,77) | -0.871 [-1.916 to 0.174] | -2.507 [-3.783 to -1.231]
  Second-Line PD: SWB (n=80,75) | -0.106 [-0.902 to 0.690] | -0.766 [-1.788 to 0.256]
  Second-Line PD: EWB (n=80,76) | -0.440 [-1.553 to 0.673] | -0.508 [-1.562 to 0.546]
  Second-Line PD: FWB (n=80,76) | -1.415 [-2.590 to -0.239] | -0.773 [-1.809 to 0.263]
  Second-Line PD: Breast Cancer (n=77,77) | 0.120 [-1.182 to 1.421] | 0.241 [-0.878 to 1.360]
  Second-Line PD: FACT-B TOI (n=74,76) | -2.311 [-5.070 to 0.447] | -3.003 [-5.734 to -0.273]
  Second-Line PD: Total FACT-G (n=76,74) | -2.771 [-5.902 to 0.361] | -4.702 [-7.941 to -1.462]
  Second-Line PD: Total FACT-B (n=72,74) | -2.719 [-6.633 to 1.195] | -4.440 [-8.515 to -0.366]

25. Primary Outcome: Percentage of Participants Estimated to be Alive and Free of Second-Line Disease Progression at Month 12
Description: Second-line PFS was defined as the time from randomization to PD or death due to any cause during their second-line of treatment with bevacizumab and/or chemotherapy, whichever occurred first. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without secondline PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: Month 12
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 16.9 [12.3 to 22.2] | 24.2 [19.0 to 29.9]

26. Primary Outcome: Percentage of Participants Estimated to be Alive and Free of Second-Line Disease Progression at Month 18
Description: Second-line PFS was defined as the time from randomization to PD or death due to any cause during their secondline of treatment with bevacizumab and/or chemotherapy, whichever occurred first. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without second-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: Month 18
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 9.9 [6.4 to 14.3] | 11.0 [7.4 to 15.5]

27. Primary Outcome: Percentage of Participants Estimated to be Alive and Free of Second-Line Disease Progression at Month 24
Description: as for outcome 14
Time Frame: Month 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CT Arm | CT+BV Arm
Number analyzed (Participants) | 247 | 247
percentage of participants | 6.4 [3.6 to 10.2] | 6.5 [3.7 to 10.2]

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 4 years.
Description: All randomized participants who received at least 1 dose of bevacizumab and/or chemotherapy were included in the analysis.
Arm/Group | CT Arm | CT+BV Arm
Serious Adverse Events (participants affected / at risk) | 55/238 | 89/245
Other Adverse Events (participants affected / at risk) | 181/238 | 218/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT Arm (N=238) | CT+BV Arm (N=245)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 12
Neutropenia (Blood and lymphatic system disorders) | 6 | 10
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Infection (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Injection site infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 2 | 4
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 1 | 2
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Device failure (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 3
Pain (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ischaemic stoke (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardiotoxicity (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Embolism venous (Vascular disorders) | 1 | 3
Haemorrhage (Vascular disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Postrenal failure (Renal and urinary disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Salpingo-oophorectomy (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Biopsy liver (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Patient-device incompatibility (General disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Large intestine anastomosis (Surgical and medical procedures) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT Arm (N=238) | CT+BV Arm (N=245)
Proteinuria (Renal and urinary disorders) | 70 | 133
Hypertension (Vascular disorders) | 55 | 90
Haemorrhage (Vascular disorders) | 7 | 29
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 58 | 72
Neutropenia (Blood and lymphatic system disorders) | 55 | 64
Leukopenia (Blood and lymphatic system disorders) | 18 | 30
Anaemia (Blood and lymphatic system disorders) | 13 | 22
Diarrhoea (Gastrointestinal disorders) | 27 | 35
Nausea (Gastrointestinal disorders) | 31 | 33
Vomiting (Gastrointestinal disorders) | 22 | 16
Fatigue (General disorders) | 33 | 49
Mucosal inflammation (General disorders) | 9 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 16
Abdominal pain (Gastrointestinal disorders) | 3 | 15
Constipation (Gastrointestinal disorders) | 9 | 13
Asthenia (General disorders) | 5 | 14
Pyrexia (General disorders) | 11 | 14
Urinary tract infection (Infections and infestations) | 2 | 16
Decreased appetite (Metabolism and nutrition disorders) | 4 | 21
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.